CLINICAL TRIAL: NCT02669836
Title: Posterior Fossa Decompression With or Without Duraplasty for Chiari Type I Malformation With Syringomyelia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Johns Hopkins All Children's Hospital (Other); Arkansas Children's Hospital Research Institute (Other); Boston Children's Hospital (Other); Children's Healthcare of Atlanta (Other); Dartmouth-Hitchcock Medical Center (Other); Children's Hospital Colorado (Other); Birmingham Children's Hospital (Other); Morgan Stanley Children's Hospital (Other); Phoenix Children's Hospital (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Children's National Research Institute (Other); Children's Hospital of Philadelphia (Other); Children's Hospital Medical Center, Cincinnati (Other); Columbia University (Other); Gillette Children's Specialty Healthcare (Other); Levine Children's Hospital (Other); Children's Hospital Los Angeles (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Mayo Clinic (Other); Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other); Medical University of South Carolina Shawn Jenkins Children's Hospital (Other); Oregon Health and Science University (Other); Penn State University (Other); University of Pittsburgh (Other); Primary Children's Hospital (Other); Seattle Children's Hospital (Other); Stanford University (Other); Baylor College of Medicine (Other); The Children's Hospital at OU Medical Center (Other); Nationwide Children's Hospital (Other); University of California (Other); University of Iowa (Other); University of Michigan (Other); The University of Texas Health Science Center, Houston (Other); University of Minnesota (Other); University of Vermont (Other); UVA Children's Hospital (Other); University of Wisconsin, Madison (Other); Vanderbilt University (Other); Wake Forest University (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCORI275- 201604044
Record Dates: First submitted 2016-01-13; First posted 2016-02-01 (Estimated); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-08

CONDITIONS: Arnold-Chiari Malformation, Type 1; Chiari Malformation Type I; Type I Arnold-Chiari Malformation; Syringomyelia
MeSH Terms: conditions — Arnold-Chiari Malformation; Syringomyelia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Posterior fossa decompression surgery (Experimental): The bone is surgically removed from the suboccipital region of the skull and Cervical 1 lamina so the constricting epidural band can be resected
  Interventions: Procedure: Posterior fossa decompression
- Dural augmentation surgery (Experimental): The bone is removed from the suboccipital region of the skull and Cervical 1 lamina so the constricting epidural band can be resected. Then, the dura is opened. Microsurgical dissection is performed and the dura is sewn closed.
  Interventions: Procedure: Dural Augmentation

INTERVENTIONS:
Procedure: Posterior fossa decompression — Planned areas of bone removal from the suboccipital region of the skull and cervical l1 lamina. Then, the constricting epidural band at the level of the foramen magnum is resected.
  Other Names: Bone only posterior decompression; Extradural posterior decompression
  Arms: Posterior fossa decompression surgery
Procedure: Dural Augmentation — The dura is opened sharply, exposing the cerebellar tonsils, brainstem, and upper spinal cord. After microsurgical dissection, the dura is sewn closed with a dural graft.
  Arms: Dural augmentation surgery

SUMMARY:
The purpose of this study is to determine whether a posterior fossa decompression or a posterior fossa decompression with duraplasty results in better patient outcomes with fewer complications and improved quality of life in those who have Chiari malformation type I and syringomyelia.

DETAILED DESCRIPTION:
Participants with Chiari Malformation type I and syringomyelia will be randomized to either have a posterior fossa decompression done with or without duraplasty. The participant will then return to the neurosurgeon's office at the following time points which are consistent with standard of care practice: < 6 weeks, 3-6 months, and 12 months. At these visits, the clinician will complete a physical exam and the participant will report on the prognosis of symptoms and complete two quality of life questionnaires. A brain and cervical spine MRI will be performed 12 months after the decompression.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤21 years old
2. Chiari malformation type I ≥5 mm tonsillar ectopia
3. Syrinx between 3 mm and 6 mm
4. Chiari Severity Index (CSI) classification 1
5. MRI of the brain and cervical and thoracic spine are required prior to surgery and must be available to be shared with the Data Coordinating Center

Exclusion Criteria:

1. CSI-2 or CSI-3 classification
2. Syrinx <3 mm and/or ≥6 mm
3. Neuro-imaging demonstrating basilar invagination
4. Clival canal angle <120° (signs of severe craniovertebral junction disease)
5. Chiari Malformation I + syringomyelia secondary to other pathology (e.g. a tumor)
6. Unable to share pre-decompression MRI of the brain and cervical and thoracic spine
7. Patients who do not wish to participate

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 162 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David D Limbrick, MD, PhD, Principal Investigator — Washington University-St. Louis Children's Hospital
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Di Lorenzo N, Cacciola F. Adult syringomielia. Classification, pathogenesis and therapeutic approaches. J Neurosurg Sci. 2005 Sep;49(3):65-72. PMID 16288188
- [Background] Heiss JD, Patronas N, DeVroom HL, Shawker T, Ennis R, Kammerer W, Eidsath A, Talbot T, Morris J, Eskioglu E, Oldfield EH. Elucidating the pathophysiology of syringomyelia. J Neurosurg. 1999 Oct;91(4):553-62. doi: 10.3171/jns.1999.91.4.0553. PMID 10507374
- [Background] Small JA, Sheridan PH. Research priorities for syringomyelia: a National Institute of Neurological Disorders and Stroke workshop summary. Neurology. 1996 Feb;46(2):577-82. doi: 10.1212/wnl.46.2.577. No abstract available. PMID 8614541
- [Background] Brickell KL, Anderson NE, Charleston AJ, Hope JK, Bok AP, Barber PA. Ethnic differences in syringomyelia in New Zealand. J Neurol Neurosurg Psychiatry. 2006 Aug;77(8):989-91. doi: 10.1136/jnnp.2005.081240. Epub 2006 Mar 20. PMID 16549414
- [Background] Arnautovic A, Splavski B, Boop FA, Arnautovic KI. Pediatric and adult Chiari malformation Type I surgical series 1965-2013: a review of demographics, operative treatment, and outcomes. J Neurosurg Pediatr. 2015 Feb;15(2):161-77. doi: 10.3171/2014.10.PEDS14295. Epub 2014 Dec 5. PMID 25479580
- [Background] Fernandez AA, Guerrero AI, Martinez MI, Vazquez ME, Fernandez JB, Chesa i Octavio E, Labrado Jde L, Silva ME, de Araoz MF, Garcia-Ramos R, Ribes MG, Gomez C, Valdivia JI, Valbuena RN, Ramon JR. Malformations of the craniocervical junction (Chiari type I and syringomyelia: classification, diagnosis and treatment). BMC Musculoskelet Disord. 2009 Dec 17;10 Suppl 1(Suppl 1):S1. doi: 10.1186/1471-2474-10-S1-S1. PMID 20018097
- [Background] Hida K, Iwasaki Y, Koyanagi I, Abe H. Pediatric syringomyelia with chiari malformation: its clinical characteristics and surgical outcomes. Surg Neurol. 1999 Apr;51(4):383-90; discussion 390-1. doi: 10.1016/s0090-3019(98)00088-3. PMID 10199291
- [Background] Mueller D, Oro' JJ. Prospective analysis of self-perceived quality of life before and after posterior fossa decompression in 112 patients with Chiari malformation with or without syringomyelia. Neurosurg Focus. 2005 Feb 15;18(2):ECP2. doi: 10.3171/foc.2005.18.2.11. PMID 15715455
- [Background] Tisell M, Wallskog J, Linde M. Long-term outcome after surgery for Chiari I malformation. Acta Neurol Scand. 2009 Nov;120(5):295-9. doi: 10.1111/j.1600-0404.2009.01183.x. Epub 2009 Jun 11. PMID 19519678
- [Background] Greenberg JK, Yarbrough CK, Radmanesh A, Godzik J, Yu M, Jeffe DB, Smyth MD, Park TS, Piccirillo JF, Limbrick DD. The Chiari Severity Index: a preoperative grading system for Chiari malformation type 1. Neurosurgery. 2015 Mar;76(3):279-85; discussion 285. doi: 10.1227/NEU.0000000000000608. PMID 25584956
- [Background] Vakharia VN, Guilfoyle MR, Laing RJ. Prospective study of outcome of foramen magnum decompressions in patients with syrinx and non-syrinx associated Chiari malformations. Br J Neurosurg. 2012 Feb;26(1):7-11. doi: 10.3109/02688697.2011.578771. Epub 2011 May 18. PMID 21591857
- [Background] Munshi I, Frim D, Stine-Reyes R, Weir BK, Hekmatpanah J, Brown F. Effects of posterior fossa decompression with and without duraplasty on Chiari malformation-associated hydromyelia. Neurosurgery. 2000 Jun;46(6):1384-9; discussion 1389-90. doi: 10.1097/00006123-200006000-00018. PMID 10834643
- [Background] Ventureyra EC, Aziz HA, Vassilyadi M. The role of cine flow MRI in children with Chiari I malformation. Childs Nerv Syst. 2003 Feb;19(2):109-13. doi: 10.1007/s00381-002-0701-1. Epub 2003 Jan 30. PMID 12607030
- [Background] Navarro R, Olavarria G, Seshadri R, Gonzales-Portillo G, McLone DG, Tomita T. Surgical results of posterior fossa decompression for patients with Chiari I malformation. Childs Nerv Syst. 2004 May;20(5):349-56. doi: 10.1007/s00381-003-0883-1. Epub 2004 Mar 12. PMID 15022006
- [Background] Limonadi FM, Selden NR. Dura-splitting decompression of the craniocervical junction: reduced operative time, hospital stay, and cost with equivalent early outcome. J Neurosurg. 2004 Nov;101(2 Suppl):184-8. doi: 10.3171/ped.2004.101.2.0184. PMID 15835106
- [Background] Yeh DD, Koch B, Crone KR. Intraoperative ultrasonography used to determine the extent of surgery necessary during posterior fossa decompression in children with Chiari malformation type I. J Neurosurg. 2006 Jul;105(1 Suppl):26-32. doi: 10.3171/ped.2006.105.1.26. PMID 16871867
- [Background] Galarza M, Sood S, Ham S. Relevance of surgical strategies for the management of pediatric Chiari type I malformation. Childs Nerv Syst. 2007 Jun;23(6):691-6. doi: 10.1007/s00381-007-0297-6. Epub 2007 Jan 25. PMID 17252266
- [Background] Mutchnick IS, Janjua RM, Moeller K, Moriarty TM. Decompression of Chiari malformation with and without duraplasty: morbidity versus recurrence. J Neurosurg Pediatr. 2010 May;5(5):474-8. doi: 10.3171/2010.1.PEDS09218. PMID 20433261
- [Background] Litvack ZN, Lindsay RA, Selden NR. Dura splitting decompression for Chiari I malformation in pediatric patients: clinical outcomes, healthcare costs, and resource utilization. Neurosurgery. 2013 Jun;72(6):922-8; discussion 928-9. doi: 10.1227/NEU.0b013e31828ca1ed. PMID 23426152
- [Background] Lee A, Yarbrough CK, Greenberg JK, Barber J, Limbrick DD, Smyth MD. Comparison of posterior fossa decompression with or without duraplasty in children with Type I Chiari malformation. Childs Nerv Syst. 2014 Aug;30(8):1419-24. doi: 10.1007/s00381-014-2424-5. Epub 2014 Apr 29. PMID 24777296
- [Background] Rocque BG, George TM, Kestle J, Iskandar BJ. Treatment practices for Chiari malformation type I with syringomyelia: results of a survey of the American Society of Pediatric Neurosurgeons. J Neurosurg Pediatr. 2011 Nov;8(5):430-7. doi: 10.3171/2011.8.PEDS10427. PMID 22044364
- [Background] Batzdorf U. Primary spinal syringomyelia. Invited submission from the joint section meeting on disorders of the spine and peripheral nerves, March 2005. J Neurosurg Spine. 2005 Dec;3(6):429-35. doi: 10.3171/spi.2005.3.6.0429. PMID 16381204
- [Background] Tubbs RS, Lyerly MJ, Loukas M, Shoja MM, Oakes WJ. The pediatric Chiari I malformation: a review. Childs Nerv Syst. 2007 Nov;23(11):1239-50. doi: 10.1007/s00381-007-0428-0. Epub 2007 Jul 18. PMID 17639419
- [Background] Wellons JC & Smyth MD (2013) Neurosurgical Face Off: Durotomy and Duraplasty Versus No Durotomy and Duraplasty. Annual Scientific Meeting of the American Association of Neurological Surgeons.
- [Background] Greenberg JK, Milner E, Yarbrough CK, Lipsey K, Piccirillo JF, Smyth MD, Park TS, Limbrick DD Jr. Outcome methods used in clinical studies of Chiari malformation Type I: a systematic review. J Neurosurg. 2015 Feb;122(2):262-72. doi: 10.3171/2014.9.JNS14406. Epub 2014 Nov 7. PMID 25380104
- [Background] Durham SR, Fjeld-Olenec K. Comparison of posterior fossa decompression with and without duraplasty for the surgical treatment of Chiari malformation Type I in pediatric patients: a meta-analysis. J Neurosurg Pediatr. 2008 Jul;2(1):42-9. doi: 10.3171/PED/2008/2/7/042. PMID 18590394
- [Background] Ladner TR, Westrick AC, Wellons JC 3rd, Shannon CN. Health-related quality of life in pediatric Chiari Type I malformation: the Chiari Health Index for Pediatrics. J Neurosurg Pediatr. 2016 Jan;17(1):76-85. doi: 10.3171/2015.5.PEDS1513. Epub 2015 Oct 2. PMID 26431245
- [Background] Guyatt GH, Kirshner B, Jaeschke R. Measuring health status: what are the necessary measurement properties? J Clin Epidemiol. 1992 Dec;45(12):1341-5. doi: 10.1016/0895-4356(92)90194-r. PMID 1460470
- [Background] Kirshner B, Guyatt G. A methodological framework for assessing health indices. J Chronic Dis. 1985;38(1):27-36. doi: 10.1016/0021-9681(85)90005-0. PMID 3972947
- [Background] Carmines EG & Zeller RA (1979) Reliability and Validity Assessment. Quatitative Applications in the Social Sciences. (Sage Publications, Newbury Park, CA).
- [Background] Feudtner C, Hays RM, Haynes G, Geyer JR, Neff JM, Koepsell TD. Deaths attributed to pediatric complex chronic conditions: national trends and implications for supportive care services. Pediatrics. 2001 Jun;107(6):E99. doi: 10.1542/peds.107.6.e99. PMID 11389297
- [Background] Yarbrough CK, Greenberg JK, Smyth MD, Leonard JR, Park TS, Limbrick DD Jr. External validation of the Chicago Chiari Outcome Scale. J Neurosurg Pediatr. 2014 Jun;13(6):679-84. doi: 10.3171/2014.3.PEDS13503. Epub 2014 Apr 11. PMID 24724715
- [Background] Weinstein JN, Lurie JD, Tosteson TD, Skinner JS, Hanscom B, Tosteson AN, Herkowitz H, Fischgrund J, Cammisa FP, Albert T, Deyo RA. Surgical vs nonoperative treatment for lumbar disk herniation: the Spine Patient Outcomes Research Trial (SPORT) observational cohort. JAMA. 2006 Nov 22;296(20):2451-9. doi: 10.1001/jama.296.20.2451. PMID 17119141
- [Background] Drake JM, Singhal A, Kulkarni AV, DeVeber G, Cochrane DD; Canadian Pediatric Neurosurgery Study Group. Consensus definitions of complications for accurate recording and comparisons of surgical outcomes in pediatric neurosurgery. J Neurosurg Pediatr. 2012 Aug;10(2):89-95. doi: 10.3171/2012.3.PEDS11233. Epub 2012 Jun 22. PMID 22725268
- [Background] Donner A & Klar N (2000) Design and Analysis of Cluster Randomization Trials in Health Research (Arnold; Oxford University Press, New York).
- [Background] Little RJA & Rubin DB (2002) Statistical Analysis With Missing Data (Wiley, Hoboken, N.J.) Second Edition Ed.
- [Background] Buck SF (1960) A method of estimation of missing values in multivariate data suitable for use with an electronic computer. J Roy Statist Soc 22:302-306.
- [Background] Godzik J, Kelly MP, Radmanesh A, Kim D, Holekamp TF, Smyth MD, Lenke LG, Shimony JS, Park TS, Leonard J, Limbrick DD. Relationship of syrinx size and tonsillar descent to spinal deformity in Chiari malformation Type I with associated syringomyelia. J Neurosurg Pediatr. 2014 Apr;13(4):368-74. doi: 10.3171/2014.1.PEDS13105. Epub 2014 Feb 14. PMID 24527859
- [Background] Greenberg JK, et al. (2014) Population-Based Analysis of Complications Associated with Chiari Malformation Type 1 Surgery in Children. AANS/CNS Joint Section on Pediatric Neurosurgery.
- [Background] Gail M, Simon R. Testing for qualitative interactions between treatment effects and patient subsets. Biometrics. 1985 Jun;41(2):361-72. PMID 4027319
- [Background] Hankinson T, Tubbs RS, Wellons JC. Duraplasty or not? An evidence-based review of the pediatric Chiari I malformation. Childs Nerv Syst. 2011 Jan;27(1):35-40. doi: 10.1007/s00381-010-1295-7. Epub 2010 Oct 2. PMID 20890606
- [Background] Marcus DS, Archie KA, Olsen TR, Ramaratnam M. The open-source neuroimaging research enterprise. J Digit Imaging. 2007 Nov;20 Suppl 1(Suppl 1):130-8. doi: 10.1007/s10278-007-9066-z. Epub 2007 Aug 21. PMID 17710494
- [Background] Marcus DS, Olsen TR, Ramaratnam M, Buckner RL. The Extensible Neuroimaging Archive Toolkit: an informatics platform for managing, exploring, and sharing neuroimaging data. Neuroinformatics. 2007 Spring;5(1):11-34. doi: 10.1385/ni:5:1:11. PMID 17426351
- [Derived] Hale AT, Adelson PD, Albert GW, Aldana PR, Alden TD, Anderson RCE, Bauer DF, Bonfield CM, Brockmeyer DL, Chern JJ, Couture DE, Daniels DJ, Durham SR, Ellenbogen RG, Eskandari R, George TM, Grant GA, Graupman PC, Greene S, Greenfield JP, Gross NL, Guillaume DJ, Heuer GG, Iantosca M, Iskandar BJ, Jackson EM, Johnston JM, Keating RF, Leonard JR, Maher CO, Mangano FT, McComb JG, Meehan T, Menezes AH, O'Neill B, Olavarria G, Park TS, Ragheb J, Selden NR, Shah MN, Smyth MD, Stone SSD, Strahle JM, Wait SD, Wellons JC, Whitehead WE, Shannon CN, Limbrick DD; Park-Reeves Syringomyelia Research Consortium Investigators. Factors associated with syrinx size in pediatric patients treated for Chiari malformation type I and syringomyelia: a study from the Park-Reeves Syringomyelia Research Consortium. J Neurosurg Pediatr. 2020 Mar 6;25(6):629-639. doi: 10.3171/2020.1.PEDS19493. Print 2020 Jun 1. PMID 32114543

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Posterior Fossa Decompression Surgery | Dural Augmentation Surgery
Started (Based on ITT including radio-graphic only visits) | 84 | 78
3-6 Month Follow up | 60 | 63
Completed | 53 | 61
Not Completed | 31 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posterior Fossa Decompression Surgery | Dural Augmentation Surgery | Total
Number analyzed (Participants) | 84 | 78 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 80 | 74 | 154
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Note: values represent reporting by ITT, i.e. split by randomization, not necessarily treatment received
  years | 9.94 (5.59) | 10.77 (5.37) | 10.34 (5.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Note: values represent reporting by ITT, i.e. split by randomization, not necesarily treatment received
  Participants
    Female | 48 | 39 | 87
    Male | 36 | 39 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Note: values represent reporting by ITT, i.e. split by randomization, not necessarily treatment received
  Participants
    Hispanic or Latino | 6 | 9 | 15
    Not Hispanic or Latino | 78 | 69 | 147
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Note: values represent reporting by ITT, i.e. split by randomization, not necesarily treatment received
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 5 | 10 | 15
    White | 72 | 59 | 131
    More than one race | 4 | 4 | 8
    Unknown or Not Reported | 2 | 4 | 6
Size of Syringomyelia [Count of Participants; unit: Participants] — Note: values represent reporting by ITT, i.e. split by randomization, not necessarily treatment received
  Participants
    Syrinx AP Diameter (mm) 3-6 mm | 65 | 37 | 102
    Syrinx AP Diameter (mm) 7-9 mm | 19 | 41 | 60

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Surgical Complications
Description: The number of participants with complications such as: Cerebrospinal fluid (CSF)-related complications ≤6 months (e.g. CSF leak, pseudomeningocele, aseptic meningitis, infection, hydrocephalus), and the requirement for additional surgery for wound revision or CSF diversion
Time Frame: less then or equal to 6 months from decompression
Population: Note: values represent reporting by ITT, i.e. split by randomization, not necessarily treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Posterior Fossa Decompression Surgery | Dural Augmentation Surgery
Number analyzed (Participants) | 84 | 78
Participants | 8 | 10

2. Secondary Outcome: Aim 2: The Number of Patients With Clinical Improvement
Description: Number of patients who experienced improvement in clinical or neurological symptoms-such as; headaches, pain, numbness or tingling, nausea/ vomiting, itching, weakness, difficulty swallowing, difficulty sleeping and cranial nerve assessments.
Time Frame: 10-14 months
Population: Note: values represent reporting by ITT, i.e. split by randomization, not necessarily treatment received
Measure: Count of Participants; unit: Participants
Arm/Group | Posterior Fossa Decompression Surgery | Dural Augmentation Surgery
Number analyzed (Participants) | 53 | 61
Participants | 43 | 43

3. Secondary Outcome: Aim 2: The Mean Number of Syrinx Reduction in Millimeters Less Than 24 Months Post Surgery.
Description: Syrinx regression comparison between posterior fossa decompression surgery and dural augmentation surgery cohorts based on ITT.
Time Frame: 10-14 months
Population: Values represent reporting by ITT not treatment received
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Posterior Fossa Decompression Surgery | Dural Augmentation Surgery
Number analyzed (Participants) | 52 | 60
millimeters | 1.06 (1.73) | 3.07 (2.47)

4. Other Pre Specified Outcome: Aim 3 : Mean Change in Quality of Life Measurement After Surgery Relative to Baseline.
Description: Quality of Life (QOL) was assessed using the Chiari Health Index Pediatrics (CHIP), and the Health Utilities-3 (HUI-3). The CHIP is a 5-point response scale. Within the physical symptoms' domain, 5 questions regarding pain severity are alternatively scaled.
  The Health Utilities Index Mark 3 (HUI3) is a generic status classification system, generalizable in pediatric patients with illness. The HUI3 assesses domains including vision, hearing, speech, ambulation, dexterity, emotion, cognition, and pain.
  We used a non-inferiority approach in the analysis. The score is corrected for missing values and scaled to a range of scores between 0 and 1. An increasing score represents increasing HRQOL. Increase/decrease in the quality of life metric (on a scale from 0-1, with 0 representing no quality of life and 1 representing 100% quality of life).
Time Frame: 10-14 Months from Decompression
Population: Note: values represent reporting by ITT, i.e. split by randomization, not necessarily treatment received
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Posterior Fossa Decompression Surgery | Dural Augmentation Surgery
Number analyzed (Participants) | 28 | 29
score on a scale | 0.02 (0.16) | 0.04 (0.17)

ADVERSE EVENTS:
Time Frame: < 6 weeks, 3-6 months and 10-14 months
Description: Patients were followed by their physician at <6 weeks, 3-6 months and 10-14 months or as needed per standard clinical care. If individuals experienced adverse events they would have been reported during those interactions.
Arm/Group | Posterior Fossa Decompression Surgery | Dural Augmentation Surgery
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/78
Other Adverse Events (participants affected / at risk) | 0/84 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT02669836/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT02669836/SAP_001.pdf